CLINICAL TRIAL: NCT07353671
Title: A Single-Center, Two-Arm, Prospective Clinical Study Evaluating the Efficacy and Safety of a Topical Periplaneta Americana-Derived Regenerative Solution (Meilian Fuxin Liquid) for the Treatment of Radiation Dermatitis
Brief Title: Topical Periplaneta Americana-Derived Meilian Fuxin Liquid for Radiation Dermatitis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025(1723)
Record Dates: First submitted 2025-12-14; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Radiation-induced Dermatitis
Keywords: Head & neck cancer; Radiation-induced Dermatitis; Meilian Fuxin Solution
MeSH Terms: conditions — Radiodermatitis; Head and Neck Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meilian Fuxin Solution (Experimental): Topical application of Periplaneta americana-derived Meilian Fuxin Solution
  Interventions: Drug: Topical application of Periplaneta americana-derived Meilian Fuxin Solution; Radiation: Radiotherapy
- Control group (Placebo Comparator): Topical application of placebo
  Interventions: Other: Topical application of placebo; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Topical application of Periplaneta americana-derived Meilian Fuxin Solution — A topical formulation derived from Periplaneta americana (Meilian Fuxin Solution).
  Other Names: MLFX; Periplaneta Americana Extract; Meilian Fuxin Ye
  Arms: Meilian Fuxin Solution
Other: Topical application of placebo — The placebo topical formulation will be composed of inactive ingredients and will be matched in appearance, texture, and administration regimen to the active Periplaneta americana-derived Meilian Fuxin Solution, and participants will also receive standard skin care for radiation dermatitis according to institutional clinical practice guidelines.
  Arms: Control group
Radiation: Radiotherapy — One of the inclusion criteria for the study was that patients with squamous carcinoma of the head and neck (including nasopharyngeal carcinoma) needed to receive either radiotherapy alone or simultaneous radiotherapy and chemotherapy.

SUMMARY:
To evaluate the efficacy and safety of topical Periplaneta americana-derived Meilian Fuxin Solution for the prevention of radiation dermatitis in patients undergoing radiotherapy.

DETAILED DESCRIPTION:
The clinical trial aims to evaluate the efficacy and safety of topical Periplaneta americana-derived Meilian Fuxin Solution in preventing and reducing radiation dermatitis in patients undergoing radiotherapy. Participants will be assigned to receive either topical Meilian Fuxin Solution or a placebo formulation, applied twice daily to the irradiated skin area from the start of radiotherapy through completion of treatment. The placebo will be administered using an identical application regimen. Radiation dermatitis will be assessed at baseline and at regular intervals during and after radiotherapy using the Radiation Therapy Oncology Group (RTOG) criteria, and safety will be evaluated by monitoring local and systemic adverse events throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Age and Gender: Patients aged 18 to 80 years (inclusive of boundary values), regardless of gender.
2. Diagnosis and Treatment: Patients with head and neck cancer (including nasopharyngeal carcinoma) who have been confirmed by histopathology and require radical radiotherapy or postoperative adjuvant radiotherapy.
3. Performance Status: Patients with an ECOG Performance Status score of 0 to 2.
4. Consent: Patients who voluntarily agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Prior Radiotherapy: Patients with a history of prior radiotherapy to the target area.
2. Baseline Skin Condition: Baseline skin condition in the treatment area that may interfere with efficacy assessment (e.g., presence of open wounds, infection, rash, psoriasis, etc.).
3. Systemic Diseases: Presence of connective tissue diseases or other systemic dermatoses.
4. Known Allergies: Known allergy to any component of the investigational product (Meilian Fuxin Solution).
5. Prior Clinical Research: Participation in other interventional clinical studies within the past 3 months and use of any investigational drugs or devices.
6. Investigator Discretion: Subjects judged by the investigator to be unsuitable for participation in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 2 or Higher Acute Radiation Dermatitis (RTOG Criteria) | The evaluation period is approximately 14 weeks to 14.5 weeks.
  Acute radiation dermatitis is assessed by trained radiation oncologists according to the Radiation Therapy Oncology Group (RTOG) acute radiation morbidity scoring criteria. The RTOG grading system categorizes acute radiation dermatitis into grades 0 to 4, with higher grades indicating more severe skin reactions. Grade 0 indicates no visible skin changes; Grade 1 indicates faint erythema or dry desquamation; Grade 2 indicates moderate to brisk erythema or patchy moist desquamation, mainly confined to skin folds; Grade 3 indicates confluent moist desquamation outside of skin folds or bleeding induced by minor trauma; and Grade 4 indicates skin necrosis or ulceration of full-thickness dermis, or spontaneous bleeding. The incidence of Grade 2 or higher acute radiation dermatitis is defined as the proportion of participants who develop Grade 2, Grade 3, or Grade 4 dermatitis at any time during radiotherapy or within the post-radiotherapy follow-up period.

SECONDARY OUTCOMES:
Incidence of Grade 3 or Grade 4 Radiation Dermatitis | The evaluation period is approximately 14 weeks and 14.5 weeks.
  Radiation dermatitis is assessed by trained physicians according to the Radiation Therapy Oncology Group (RTOG) acute radiation morbidity scoring criteria.
Time to Occurrence of Grade 3 or Grade 4 Radiation Dermatitis | The evaluation period is approximately 14 weeks to 14.5 weeks.
  The time from the start of radiotherapy to the first documented occurrence of Grade 3 or Grade 4 radiation dermatitis, as assessed according to the Radiation Therapy Oncology Group (RTOG) acute radiation morbidity scoring criteria.
The duration of any-grade Radiation Dermatitis | The evaluation period is approximately 14 weeks and 14.5 weeks.
  The first determination of radiation dermatitis to the first instance of non-radiation dermatitis, without a subsequent instance of radiation dermatitis.
Change in Radiation Dermatitis Severity Score using the RISRAS Scale | The evaluation period is approximately 14 weeks and 14.5 weeks.
  The change in radiation dermatitis severity, as measured by the Radiation-Induced Skin Reaction Assessment Scale (RISRAS), which ranges from 0 to 24, with higher scores indicating more severe skin reactions. Scores will be assessed at baseline (before the first day of radiotherapy), weekly during radiotherapy, and at follow-up visits up to 8 weeks after completion of radiotherapy.
Change in Patient Quality of Life using the Skindex-16 | The evaluation period is approximately 14 weeks and 14.5 weeks.
  The change in patient-reported quality of life related to skin symptoms, as measured by the Skindex-16 Dermatology Life Quality Instrument, which ranges from 0 to 100, with higher scores indicating worse quality of life. Scores will be assessed at baseline (before the first day of radiotherapy), weekly during radiotherapy, and at follow-up visits up to 8 weeks after completion of radiotherapy.
Radiotherapy Interruption due to Radiation Dermatitis | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6.5 weeks.
  The occurrence of any temporary interruption, delay, or discontinuation of radiotherapy attributable to radiation dermatitis, as documented in the medical record. The reason for interruption will be confirmed by the treating radiation oncologist.
Adverse events | The evaluation period is approximately 14 weeks and 14.5 weeks.
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version

OTHER OUTCOMES:
Overall Health Status and Core Dimensions of Quality of Life | The total evaluation period is approximately 14 to 14.5 weeks.
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) This instrument is a 30-item patient-reported outcome (PRO) measure designed to evaluate core aspects of health-related quality of life in cancer patients, including 5 functional scales (physical, role, cognitive, emotional, social), 3 symptom scales (fatigue, pain, nausea and vomiting), one global health status/quality of life scale, and 6 single-item symptom measures. Scores are linearly transformed to a range of 0-100. For the functional scales and the global health status scale, higher scores indicate better functional levels or quality of life; for the symptom scales/items, higher scores indicate greater symptom burden.
Head and Neck Cancer-Specific Symptoms | The total evaluation period is approximately 14 to 14.5 weeks.
  The EORTC QLQ-H&N35 is a patient-reported outcome (PRO) instrument specifically designed to assess disease-related symptoms and treatment-related side effects in patients with head and neck cancer. It comprises 35 items, organized into seven multi-item subscales (pain, swallowing, senses, speech, social eating, social contact, and sexuality) and eleven single-item measures (such as dental problems, problems opening mouth, sticky saliva, coughing, etc.). All subscale and single-item scores are linearly transformed to a 0-100 scale using a standardized scoring algorithm. Interpretation of Scores: For all subscales and single items, higher scores represent more severe symptoms or greater symptom burden.
The number of patients who missed five or more consecutive radiation fractions | The evaluation period is approximately 6 weeks and 6.5 weeks.
  The number of patients who missed five or more consecutive radiations and the reasons for this are recorded during radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — West China Hospital
Locations (1):
- Sichuan University West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No